CLINICAL TRIAL: NCT06200883
Title: Effects of a Nutraceutic Compound on Cognitive Impairment in Frailty Patients
Brief Title: Effects of a Nutraceutic Compound on Cognitive Impairment
Acronym: ENUCCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, RAFFAELE IZZO, Raffaele Izzo, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEREBRAIN
Record Dates: First submitted 2023-12-21; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Physical frailty; Cognitive frailty; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo oral tablet. In the Placebo group the participants take vehicle (1 vial per os every 24 hours) for 4 weeks
  Interventions: Drug: Placebo oral vial
- CERBRAIN (Active Comparator): In the CEREBRAIN group the participants take CEREBRAIN (1 vial per os of 1.2 g every 24 hours) for 4 weeks
  Interventions: Drug: Choline Bitartrate

INTERVENTIONS:
Drug: Placebo oral vial — In the Placebo group the participants take vehicle (1 vial per os every 24 hours) for 4 weeks
  Arms: Placebo
Drug: Choline Bitartrate — In the CEREBRAIN group the participants take CEREBRAIN (1 vial per os of 1.2 g every 24 hours) for 4 weeks
  Arms: CERBRAIN

SUMMARY:
The study is designed to evaluate the effects of choline bitartrate on cognitive impairment in frailty patients.

The study will analyze the impact of 4 weeks treatment randomized with a nutraceutical compound in a double-blind randomized placebo controlled trial. The investigators will also assess cognitive frailty.

DETAILED DESCRIPTION:
The patients and controls will be recruited at the Hypertension research center of Federico II university hospital.

The overall duration of the study will be 4 weeks for each participant. Blood pressure, heart rate and cognitive frailty and cognitive impairment will be evaluated for each patient at randomization and after 4 weeks of treatment.

Patients or controls will be randomized to receive the nutraceutical compound (1 vial of CEREBRAIN per os with 1200 mg of choline bitartrate every 24 hours) or placebo (1 vial per os without active substance every 24 hours). Before the start of treatment, patients will undergo full examination of cognitive functions (MoCA and MMSE tests, the parameters will be reported in a password-protected database, using a identification code. The duration of the treatment will be 4 weeks. At the end of the treatment, the patients will repeat the tests and the results will be identified through the use of an alphanumeric code (POST-XXXYYY).

All CEREBRAIN and placebo, made up of the CEREBRAIN vehicle without the active substance, will be offered free of charge by the Farmaceutici DAMOR company.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment

Exclusion Criteria:

Ictus Atrial fibrillation Kidney diseases Cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive functions | 4 weeks
  Cognitive functions will be assessed by MoCA test
Change in Cognitive functions | 4 weeks
  Cognitive functions will be assessed by MMSE test

SECONDARY OUTCOMES:
Change in cognitive frailty | 4 weeks
  Cognitive frailty will be assessed by the Fried criteria (at least 3/5 criteria whether MCI is diagnosed with the Clinical Dementia Rating Scale (0 to 5)

CONTACTS AND LOCATIONS:
Locations (1):
- Ambulatorio Ipertensione e Unità Coronarica Federico II University, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calabrese C, Gregory WL, Leo M, Kraemer D, Bone K, Oken B. Effects of a standardized Bacopa monnieri extract on cognitive performance, anxiety, and depression in the elderly: a randomized, double-blind, placebo-controlled trial. J Altern Complement Med. 2008 Jul;14(6):707-13. doi: 10.1089/acm.2008.0018. PMID 18611150
- [Result] Cenacchi T, Bertoldin T, Farina C, Fiori MG, Crepaldi G. Cognitive decline in the elderly: a double-blind, placebo-controlled multicenter study on efficacy of phosphatidylserine administration. Aging (Milano). 1993 Apr;5(2):123-33. doi: 10.1007/BF03324139. PMID 8323999
- [Result] Kesse-Guyot E, Fezeu L, Andreeva VA, Touvier M, Scalbert A, Hercberg S, Galan P. Total and specific polyphenol intakes in midlife are associated with cognitive function measured 13 years later. J Nutr. 2012 Jan;142(1):76-83. doi: 10.3945/jn.111.144428. Epub 2011 Nov 16. PMID 22090468
- [Result] Kuriyama S, Hozawa A, Ohmori K, Shimazu T, Matsui T, Ebihara S, Awata S, Nagatomi R, Arai H, Tsuji I. Green tea consumption and cognitive function: a cross-sectional study from the Tsurugaya Project 1. Am J Clin Nutr. 2006 Feb;83(2):355-61. doi: 10.1093/ajcn/83.2.355. PMID 16469995
- [Result] Mastroiacovo D, Kwik-Uribe C, Grassi D, Necozione S, Raffaele A, Pistacchio L, Righetti R, Bocale R, Lechiara MC, Marini C, Ferri C, Desideri G. Cocoa flavanol consumption improves cognitive function, blood pressure control, and metabolic profile in elderly subjects: the Cocoa, Cognition, and Aging (CoCoA) Study--a randomized controlled trial. Am J Clin Nutr. 2015 Mar;101(3):538-48. doi: 10.3945/ajcn.114.092189. Epub 2014 Dec 17. PMID 25733639
- [Result] Mohamed S, Lee Ming T, Jaffri JM. Cognitive enhancement and neuroprotection by catechin-rich oil palm leaf extract supplement. J Sci Food Agric. 2013 Mar 15;93(4):819-27. doi: 10.1002/jsfa.5802. Epub 2012 Sep 24. PMID 23001939
- [Result] Morris MC, Evans DA, Tangney CC, Bienias JL, Wilson RS. Associations of vegetable and fruit consumption with age-related cognitive change. Neurology. 2006 Oct 24;67(8):1370-6. doi: 10.1212/01.wnl.0000240224.38978.d8. PMID 17060562
- [Result] Snitz BE, O'Meara ES, Carlson MC, Arnold AM, Ives DG, Rapp SR, Saxton J, Lopez OL, Dunn LO, Sink KM, DeKosky ST; Ginkgo Evaluation of Memory (GEM) Study Investigators. Ginkgo biloba for preventing cognitive decline in older adults: a randomized trial. JAMA. 2009 Dec 23;302(24):2663-70. doi: 10.1001/jama.2009.1913. PMID 20040554